### DATA ANALYSIS PLAN

Protocol Title: A Phase 2 Randomized, Double-Blind, Placebo-

Controlled Study of ATR-101 for the Treatment of

Cushing's Syndrome

Protocol Number: ATR-101-301

Current Protocol: Global Amendment 2 / 14-MAR-2019

NCT Number: NCT03053271

Product: Nevanimibe HCl (ATR-101)

Phase of Study: 2

Sponsor: Millendo Therapeutics US, Inc.

Data Analysis Plan V1.0 / 18-SEP-2019

## <u>Protocol</u>: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of ATR-101 for the Treatment of Cushing's Syndrome

**Protocol Number:** ATR-101-301 Global Amendment 2 / 14-MAR-2019 **Current Protocol:** DAP: V1.0 / 18-SEP-2019 This Data Analysis Plan has been reviewed and approved by: Miriam Zangmeister, MS DD-MMM-YYYY Project Statistician Medpace Phillippa Miranda, MD DD-MMM-YYYY Medical Director Medpace Vivian Lin, MD DD-MMM-YYYY Vice President, Clinical Development

Millendo Therapeutics US, Inc.

## **REVISION HISTORY**

| Version | Date | Description of Changes |
|---------|-------------|-------------------------|
| 1.0 | 18-SEP-2019 | Original signed version |

## TABLE OF CONTENTS

| 1 | Intro | oduction | 5 |
|---|---|---|---|
| | 1.1 | Subject Disposition | 5 |
| | 1.2 | Demographic and Baseline Characteristics | |
| | 1.3 | 24 Hour Urinary Free Cortisol | |
| | 1.4 | Pharmacokinetics | |
| | 1.4.1 | Handling Missing Data or Concentration Below the Lower Limit of Quantification | |
| | 1.4.2 | Pharmacokinetic Parameters | |
| | 1.4.3 | Pharmacokinetic Summaries | 7 |
| | 1.5 | Adverse Events | 7 |
| | 1.6 | Clinical Safety Laboratory Evaluations | 8 |
| 2 | | les | |
| 3 | | ıres | |
| | _ | ings | |

#### 1 Introduction

This purpose of this document is to provide specifications for the tables and listings to be provided for Millendo Therapeutics Protocol ATR-101-301. Information regarding the study objectives and procedures can be found in the Protocol.

On August 12, 2019, Millendo Therapeutics elected to discontinue the ATR-101-301 study based on an analysis of the feasibility of patient recruitment and a reprioritization of resources. A total of 4 subjects entered the open-label dose-escalation period of the study, but no subjects entered the double-blind randomized withdrawal period prior to study discontinuation. The available data from subjects who participated in the study will be used for safety summaries, but no formal statistical analysis of safety data will be conducted. The efficacy parameter of 24-hour urinary free cortisol (24-hr UFC) will be summarized but formal statistical analysis will not be performed due to the limited data available.

All available data will be listed. All summaries will be based on observed values only.

#### 1.1 Subject Disposition

Counts of subjects who screened, entered the open-label dose-escalation period (i.e. dosed), and entered the double-blind randomized withdrawal period (i.e. randomized), as well as counts and percentages of subjects who completed the study and who withdrew early from the study, with the reason for early withdrawal, will be presented in total.

### 1.2 Demographic and Baseline Characteristics

Descriptive summaries of demographic and baseline characteristics will be presented for all dosed subjects. Baseline measurements refer to the last measurement prior to the first dose of study drug.

Demographic and baseline characteristics include, but are not limited to: age at informed consent, sex, race, ethnicity, height at screening, baseline body weight, and baseline body mass index (BMI). Continuous variables (age, height, weight, BMI) will be summarized by subject count, mean, standard deviation, median, minimum, and maximum. Categorical variables (race, sex, ethnicity) will be summarized by the number and percentage of subjects in the corresponding categories.

#### 1.3 24 Hour Urinary Free Cortisol

Descriptive summaries of 24-hr UFC will be presented for all dosed subjects by scheduled visit.

#### 1.4 Pharmacokinetics

Plasma PK samples will be collected to determine the concentrations of nevanimibe HCl (ATR-101; hereafter, "nevanimibe"). Planned sampling time points are listed in the table below. No subjects entered the double-blind randomized withdrawal period, therefore PK samples are not available for R1 and R2.

| Visit | Sampling Time Points (Morning Dose Only) |
|---|---|
| T1 (Day 1, 250 mg BID), | 0 (within 30 min predose), 1 (± 5 min), 2 (± 10 min), 3 (± |

| Visit | Sampling Time Points (Morning Dose Only) |
|------------------------------|------------------------------------------|
| T2 (Day 15, 500 mg) BID, and | 10 min) and 4 hr (± 10 min) |
| T3 (Day 29, 1000 mg BID) | |
| Early Termination | 0 hr |

The exact time of each sample collection will be recorded. If the exact time (measured from dosing) is outside of the collection window for nominal time points, the corresponding concentration will be excluded from concentration versus time descriptive statistical summaries and plots, but will still be used in the calculations of PK parameter estimates.

#### 1.4.1 Handling Missing Data or Concentration Below the Lower Limit of Quantification

Concentrations below the limit of quantitation (BLQ) before the first measurable concentration in a profile will be assigned a value of zero. A single BLQ value between measurable concentrations in a profile will be set to missing in the derivation of PK parameters, statistical analyses, and the individual subject plots. BLQ values that occur after the last measurable concentration will also be set to missing in the derivation of PK parameters and in the individual subject plots.

In cases of missing pre-dose at T1 visit, the missing concentrations will be assumed as zero. In cases of missing pre-dose on T2 or T3 visits, the minimum observed concentration during the dosing interval may be used as pre-dose concentration values. For other cases, the missing data will not be imputed.

#### 1.4.2 Pharmacokinetic Parameters

The following PK parameters will be estimated at T1, T2, and T3 visits for nevanimibe as data permit and as appropriate.

| PK Parameter | Definition |
|---|---|
| C <sub>max</sub> | The maximum drug concentration determined directly from individual concentration-time data |
| T <sub>max</sub> | The observed time to reach maximum concentration |
| AUC <sub>0-t</sub> | The area under the concentration-time curve from time zero to the time of the last quantified concentration |
| AUC <sub>0-4</sub> | The area under the concentration-time curve from time zero to 4 h after dosing |
| λz | The terminal phase rate constant, estimated by linear regression through the terminal phase of the log concentration-time profile |

| PK Parameter | Definition |
|---|---|
| t <sub>1/2</sub> | The terminal phase half-life, calculated as: $t\frac{1}{2} = \ln(2) \div \lambda z$ |
| $\mathrm{AUC}_{0\text{-}\infty}$ | The area under the concentration versus time curve from time 0 to infinity (first dose only), calculated as $AUC_{0-t} + C_{last}/\lambda z$ |
| AUC%extrap | Percentage of $AUC_{0-\infty}$ extrapolated, represented as $(1 - AUC_{0-t}/AUC_{0-\infty}) \times 100$ |

Plasma PK parameters will be calculated by standard non-compartmental analysis (NCA) for all dosed subjects with available data. The actual dosing and sampling time points will be used for evaluation of PK data. The linear up/log down method will be used in the computation of AUCs.

The  $\lambda z$  will not be presented for subjects who do not exhibit a terminal elimination phase in their concentration-time profiles. In order to estimate terminal elimination rate constant,  $\lambda z$ , linear regression of concentration in logarithm scale versus time will be performed using at least 3 data points. Uniform weighting will be selected to perform the regression analysis to estimate  $\lambda z$ .

Generally, the constant  $\lambda z$  will not be assigned if one of the following happens:

- 1.  $T_{\text{max}}$  is one of the 3 last data points,
- 2. The regression coefficient (R-squared) is less than 0.80,
- 3. The estimated elimination rate indicates a positive slope, or
- 4. The terminal elimination phase is not linear (as appears in a semi-logarithmic scale) based on visual inspection.

If the  $\lambda z$  is not assigned, the values of associated PK parameters will not be calculated. In the cases where AUC%extrap exceeds 20%, the  $\lambda z$  will be assigned but the  $\lambda z$  and the corresponding  $\lambda z$ -related PK parameters will be flagged and listed with an explanatory footnote.

#### 1.4.3 Pharmacokinetic Summaries

Plasma concentrations of nevanimibe will be summarized by nevanimibe dose (250 mg, 500 mg, 1000 mg) by time point, including plots in linear and semi-log scales. If the exact time (measured from dosing) is outside the collection window for the scheduled time point, the corresponding concentration is excluded from the summary of that time point.

Individual concentrations at each nevanimibe dose level will be plotted in linear and semi-log scales.

PK parameters at at each nevanimibe dose level will be summarized.

#### 1.5 Adverse Events

Adverse events (AEs) will be coded and classified by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.0. All AEs,

regardless of relationship to study drug, should be collected beginning from the time the subject signs the study consent until the last study visit or 30 days after the last dose of study drug, whichever is later. (Any SAE judged by the Investigator to be related to the study treatment should be reported to the Sponsor regardless of the length of time that has passed since study completion.) AEs in study subjects include any change in the subject's condition. This includes symptoms, physical findings, or clinical syndromes.

Treatment-emergent adverse events (TEAEs) will be defined as any adverse event beginning on or after the first dose date of study drug. AE subject counts will be provided for all dosed subjects in total and by treatment at AE onset (nevanimibe 250 mg, 500 mg, or 1000 mg).

An overview with counts of events and subjects will be provided for the incidence of AEs in the following categories.

- Any AE
- Any TEAE
- Maximum severity of TEAE
- Any study drug related TEAE
- Maximum severity of study drug related TEAE
- Any serious AE (SAE)
- AE leading to discontinuation from study drug

The incidence of TEAEs will be summarized by treatment at onset and in total by system organ class and preferred term. The same summaries will be done for study drug related TEAEs.

#### 1.6 Clinical Safety Laboratory Evaluations

Shift tables from baseline to the worst post-dose value will be presented for ALT and AST (>1xULN to 3xULN, >3xULN to 5xULN, >5xULN) and alkaline phosphatase and total bilirubin (>1xULN to 1.5xULN, >1.5xULN to 2xULN, >2xULN).

| 2 | <b>Tables</b> | |
|---|---|---|
| Tab | le 14.1.1.1 | |
| Sı | abject Disp | osition |
| | ll Subjects | |
| | | 11 |
| Sı | ummary of | Demographic and Baseline Characteristics |
| | ll Dosed Su | |
| | | 24 hour Urinary Free Cortisol |
| A | ll Dosed Su | bjects |
| | | 14 |
| | • | Pharmacokinetic Plasma Concentrations |
| A | ll Dosed Su | bjects |
| | | etic Plasma Parameter Listing and Summary |
| _ A | ll Dosed Su | bjects |
| | | Adverse Events |
| | ll Dosed Su | |
| | - | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term |
| | ll Dosed Su | |
| | - | Study Drug Related Treatment-Emergent Adverse Events by System Organ Class |
| | nd Preferred | |
| | ll Dosed Su | |
| | | falt AST Alledias Disselletons and Total Dilindia |
| | | f ALT, AST, Alkaline Phosphatase, and Total Bilirubin |
| Α | ll Dosed Su | idjecis |

## Table 14.1.1.1 Subject Disposition All Subjects

| | Total |
|--------------------------------------------------------|------------|
| Category | n (%) |
| Screened | ## |
| Entered Open-Label Dose-Escalation Period (i.e. Dosed) | 4 |
| Nevanimibe 250 mg BID | 4 (###.#) |
| Nevanimibe 500 mg BID | 4 (###.#) |
| Nevanimibe 1000 mg BID | 3 (###.#) |
| Entered Double-Blind Randomized Withdrawal Period | ## (###.#) |
| Completed the Study | ## (###.#) |
| Early termination | ## (###.#) |
| Primary reason for early termination: | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ## (###.#) |

Percentages are calculated with the number of subjects that entered the open-label dose escalation period as the denominator. Note: Subject 103-001 received nevanimibe 250 mg BID, 250 mg BID, and 500 mg BID at T1, T2, and T3 visits, respectively, instead of the planned 250 mg BID, 500 mg BID, and 1000 mg BID doses.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: Only reasons for withdrawal with total>0 will be displayed. Reasons will be sorted by descending total, then alphabetically. If reason of "other" occurs in the data, it will always appear last. >>

Protocol ATR-101-301 Page 1 of 2

#### Table 14.1.2.1 Summary of Demographic and Baseline Characteristics All Dosed Subjects

| Characteristic | Total |
|-------------------------------------------|------------|
| Category/Statistic | (N=#) |
| Age at Informed Consent | |
| n | ## |
| Mean | ##.# |
| Standard Deviation | ##.## |
| Median | ##.# |
| Minimum | ## |
| Maximum | ## |
| Sex, n (%) | |
| Female | ## (###.#) |
| Male | ## (###.#) |
| Ethnicity, n (%) | |
| Hispanic or Latino | ## (###.#) |
| Not Hispanic or Latino | ## (###.#) |
| Race, n (%) | |
| White | ## (###.#) |
| Black or African American | ## (###.#) |
| Asian | ## (###.#) |
| American Indian or Alaskan Native | ## (###.#) |
| Native Hawaiian or Other Pacific Islander | ## (###.#) |
| Multiple | ## (###.#) |

Baseline is defined as the last measurement prior to the first dose of study drug. %=100\*n/N where n is the number of subjects in the specified category and N is the number of dosed subjects.

Protocol ATR-101-301 Page 2 of 2

#### Table 14.1.2.1 Summary of Demographic and Baseline Characteristics All Dosed Subjects

| | | <del></del> |
|----------------------------------|--------|-------------|
| Characteristic | Total | |
| Category/Statistic | (N=#) | |
| Height at Screening (cm) | | |
| n | ## | |
| Mean | ##.## | |
| Standard Deviation | ##.## | |
| Median | ##.## | |
| Minimum | ##.# | |
| Maximum | ##.# | |
| Baseline Weight (kg) | | |
| n | ## | |
| Mean | ##.## | |
| Standard Deviation | ##.## | |
| Median | ##.## | |
| Minimum | ##.# | |
| Maximum | ##.# | |
| Baseline Body Mass index (kg/m²) | | |
| n | ## | |
| Mean | ##.## | |
| Standard Deviation | ##.### | |
| Median | ##.## | |
| Minimum | ##.# | |
| Maximum | ##.# | |

Baseline is defined as the last measurement prior to the first dose of study drug. %=100\*n/N where n is the number of subjects in the specified category and N is the number of dosed subjects.

Millendo Therapeutics US, Inc. Protocol ATR-101-301

Page 1 of 1

## Table 14.2.1.1 Summary of 24 hour Urinary Free Cortisol All Dosed Subjects

| Parameter (Unit)<br>Statistic | Screening | Т1 | Т2 | Т3 | ET^ | |
|---|---|---|---|---|---|---|
| XXXXXXXXX (XXXXX) | | | | | | - |
| n | 4 | 4 | 4 | 4 | 2 | |
| Mean | ##.## | ##.## | ##.## | ##.## | ##.## | |
| Standard Deviation | ##.## | ##.### | ##.### | ##.## | ##.### | |
| Median | ##.## | ##.## | ##.## | ##.## | ##.## | |
| Minimum | ##.# | ##.# | ##.# | ##.# | ##.# | |
| Maximum | ##.# | ##.# | ##.# | ##.# | ##.# | |

For Screening values, the screening collections 1 and 2 are averaged for each subject prior to summarization. The 24-hr UFC values shown are those collected after each of the indicated visits, and prior to the next visit, as follows:

^ET = End of Treatment/Early Termination Visit. Subjects 103-001 and 201-003 (both enrolled under Global Protocol Amendment 1) had 24-hr UFC summarized as occurring at ET. These collections began at Day 51 and Day 48, respectively. For 103-001, this was 8 days after last dose. For 201-003, it was the same day as last dose.

For subject 112-001, who was enrolled under Global Protocol Amendment 2, collections 1 and 2 for each timepoint are averaged prior to summarization.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< Programming Note: Source: LB.LBCAT = "24 HOUR URINE" and LBTEST = "Cortisol Excretion Rate, Free". >>

T1 = Open Label Dose Escalation Visit 1

T2 = Open Label Dose Escalation Visit 2

T3 = Open Label Dose Escalation Visit 3

# Table 14.2.2.1 Summary of Pharmacokinetic Plasma Concentrations All Dosed Subjects

| Analyte (Unit)<br>Dose Level | Scheduled<br>Time Point | N | Mean | Standard<br>Deviation | CV% | Standard<br>Error | Median | Minimum | Maximum | Geometric<br>Mean | Geometri<br>CV% |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Nevanimibe (XXXX) | | | | | | | | | | | |
| Nevanimibe 250 mg | Pre-dose | ## | #.### | #.### | ##.# | #.### | #.### | #.## | #.## | #.### | ##.# |
| - | 1 hour | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 2 hours | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 3 hours | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 4 hours | ## | #.### | #.### | ##.# | #.### | #.### | #.## | #.## | #.## | ##.# |
| Nevanimibe 500 mg | Pre-dose | ## | #.### | #.### | ##.# | #.### | #.### | #.## | #.## | #.### | ##.# |
| | 1 hour | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 2 hours | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 3 hours | ## | #.### | #.### | ##.# | #.### | #.### | #.## | #.## | #.### | ##.# |
| | 4 hours | ## | #.## | #.### | ##.# | #.### | #.### | #.## | #.## | #.## | ##.# |
| Nevanimibe 1000 mg | Pre-dose | ## | #.### | #.### | ##.# | #.### | #.### | #.## | #.## | #.### | ##.# |
| - | 1 hour | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 2 hours | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 3 hours | ## | #.### | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |
| | 4 hours | ## | # . # # # | #.### | ##.# | #.#### | #.### | #.## | #.## | #.### | ##.# |

Subjects with missing samples, below the limit of quantitation (BLQ) results that are set to missing, or samples collected out of window are not included. Geometric  $CV\% = 100*(exp(SD^2)-1)^0.5$ , where SD is the standard deviation of the log-transformed data.

## Table 14.2.2.2 Pharmacokinetic Plasma Parameter Listing and Summary All Dosed Subjects

| Analyte | Dose Level<br>Subject/Statistic | Cmax<br>(ng/mL) | Tmax<br>(h) | Lambda Z<br>(/h) | T1/2<br>(h) | AUC<br>(0-last)<br>(h*ng/mL) | AUC<br>(0-4)<br>(h*ng/mL) | AUC<br>(0-inf)<br>(h*ng/mL) | AUC%extrap<br>(%) |
|---|---|---|---|---|---|---|---|---|---|
| Nevanimibe | Nevanimibe 250 mg | | | | | | | | |
| | ###-## | ### | ##.## | #.### | ##.## | ### | ### | ### | ###.# |
| | ###-### [1] | ### | ##.## | #.### | ##.## | ### | ### | ### | ###.# |
| | ###-## | ### | ##.## | #.### | ##.## | ### | ### | ### | ###.# |
| | ###-## | ### | ##.## | #.### | ##.## | | | | |
| | n | ### | ## | # | ## | ### | ### | ### | ### |
| | Mean | ###.# | ##.## | #.### | ##.### | ###.# | ###.# | ###.# | ###.## |
| | Standard Deviation | ###.## | ##.### | #.#### | ##.### | ###.## | ###.## | ###.## | ###.### |
| | CV% | ###.# | ##.# | #.# | ##.# | ###.# | ###.# | ###.# | ###.# |
| | Standard Error | ###.## | ##.### | #.#### | ##.### | ###.## | ###.## | ###.## | ###.### |
| | Median | ###.# | ##.## | #.### | ##.### | ###.# | ###.# | ###.# | ###.## |
| | Minimum | ### | ##.## | #.### | ##.## | ### | ### | ### | ###.# |
| | Maximum | ### | ##.## | #.### | ##.## | ### | ### | ### | ###.# |
| | Geometric Mean | ###.# | N/A | N/A | N/A | ###.# | ###.# | ###.# | N/A |
| | Geometric CV% | ###.# | N/A | N/A | N/A | ###.# | ###.# | ###.# | N/A |

Geometric  $CV\%=100*(exp(SD^2)-1)^0.5$ , where SD is the standard deviation of the log-transformed data. N/A=Not Applicable.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: Repeat for each dose level. >>

<sup>[1]</sup> AUCextr > 20%, implying greater uncertainty in pharmacokinetic parameters dependent on the definition of the terminal phase and/or this extrapolation.

## Table 14.3.1.1 Overview of Adverse Events All Dosed Subjects

| | Nevanimibe Dose at Onset | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 250 mg BID<br>(N=#) | | N=#) | | 500 mg BID<br>(N=#) | | | (N=#) | | ) | | | Total (N=#) | |
| Category | n (% | | е | n | (% | ) | е | n | (%) | | е | n | (응) | е |
| Subjects with any adverse event (AE) | | | | | | | | | | | | # | (###.#) | # |
| Subjects with any treatment-emergent AE (TEAE) | # (### | #) | # | # | (### | .#) | # | # | (###. | #) | # | # | (###.#) | # |
| Maximum severity of TEAE | | | | | | | | | | | | | | |
| Mild | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Moderate | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Severe | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Subjects with any study drug related TEAE | # (### | #) | # | # | (### | .#) | # | # | (###. | #) | # | # | (###.#) | # |
| Maximum severity of study drug related TEAE | | | | | | | | | | | | | | |
| Mild | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Moderate | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Severe | # (### | #) | N/A | # | (### | .#) | N/A | # | (###. | #) | N/A | # | (###.#) | N/A |
| Subjects with any serious AE (SAE) | # (### | #) | # | # | (### | .#) | # | # | (###. | #) | # | # | (###.#) | # |
| Subjects with any AE leading to discontinuation of study drug | # (### | #) | # | # | (### | .#) | # | # | (###. | #) | # | # | (###.#) | # |

%=100\*n/N, where n is the number of subjects in the specified category and N is the number of dosed subjects per column. e = number of AEs in the specified category. AEs are summarized by the dose level at the onset of the event. TEAEs are defined as any AE beginning on or after the first dose date of study drug. Study drug related AEs include those that are possibly, probably, or definitely related.

## ${\it Table~14.3.1.2}$ Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term All Dosed Subjects

| | N | Mevanimibe Dose at | Onset | |
|---|---|---|---|---|
| System Organ Class | 250 mg BID<br>(N=#) | 500 mg BID<br>(N=#) | 1000 mg BID<br>(N=#) | Total (N=#) |
| Preferred Term | n (%) e | n (%) e | n (%) e | n (%) e |
| Subjects with any TEAE | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |
| · | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | # (###.#) # | # (###.#) # | # (###.#) # | # (###.#) # |

%=100\*n/N, where n is the number of subjects in the specified category and N is the number of dosed subjects per column. e = number of adverse events in the specified category. Treatment-emergent adverse events (TEAEs) are defined as any AE beginning on or after the first dose date of study drug. AEs are summarized by the dose level at the onset of the event. At each level of summation (overall, system organ class, preferred term), subjects reporting more than one AE are counted only once. A subject may contribute to more than one preferred term. AEs are coded using MedDRA dictionary version 18.0.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note:</u> Table will be sorted by descending frequency (n then e) in the total column for system organ class and preferred term within system organ class. >>

### << <u>Programming Note:</u> The following tables will have the same layout as Table 14.3.1.2: >>

Table 14.3.1.3

Summary of Study Drug Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term All Dosed Subjects

### << <u>Programming Note</u>: Replace

Subjects with any TEAE

With

Subjects with any study drug related TEAE

### << <u>Programming Note</u>: Include the additional footnote: >>

Study drug related AEs include those that are possibly, probably, or definitely related.

## Table 14.3.3.1 Shift Table of ALT, AST, Alkaline Phosphatase, and Total Bilirubin All Dosed Subjects

| | | Highest Post-Baseline Value | | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Normal<br>or Low<br>n (%) | >1 to<br>3xULN<br>n (%) | >3 to<br>5xULN<br>n (%) | >5xULN<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| ALT | Normal or Low | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >1 - 3xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >3 - 5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Missing | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Total | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (100.0) |
| | Normal or Low | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >1 - 3xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >3 - 5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Missing | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Total | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (100.0) |

ALT = Alanine Aminotransferase. AST = Aspartate Aminotransferase. ULN = upper limit of normal. Baseline is defined as the last measurement prior to the first dose of study drug. \$=100\*n/N, where n is the number of subjects in the specified category and N is the number of dosed subjects (N=4).

## Table 14.3.3.1 Shift Table of ALT, AST, Alkaline Phosphatase, and Total Bilirubin All Dosed Subjects

| | | Highest Post-Baseline Value | | | | | |
|---|---|---|---|---|---|---|---|
| Parameter | Baseline | Normal<br>or Low<br>n (%) | >1 to<br>1.5xULN<br>n (%) | >1.5 to<br>2xULN<br>n (%) | >2xULN<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| Alkaline Phosphatase | Normal or Low | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| marrie riiospiiasass | >1 - 1.5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >1.5 - 2xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >2xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Missing | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Total | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (100.0) |
| irubin | Normal or Low | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >1 - 1.5xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >1.5 - 2xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | >2xULN | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Missing | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) |
| | Total | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (##.#) | # (100.0) |

ALT = Alanine Aminotransferase. AST = Aspartate Aminotransferase. ULN = upper limit of normal. Baseline is defined as the last measurement prior to the first dose of study drug. \$=100\*n/N, where n is the number of subjects in the specified category and N is the number of dosed subjects (N=4).

| 3 | Figures | |
|--------|--------------------------------------|----|
| Figure | 14.2.1.1 | 22 |
| Mea | n Nevanimibe Plasma Concentrations | |
| A11 1 | Dosed Subjects | |
| Figure | 14.2.1.2 | 23 |
| Indi | vidual ATR-101 Plasma Concentrations | |
| A11 1 | Dosed Subjects | |

Figure 14.2.1.1
Mean Nevanimibe Plasma Concentrations
All Dosed Subjects



Figure 14.2.1.2
Individual ATR-101 Plasma Concentrations
All Dosed Subjects



### 4 Listings

| Listing 16.2.1.1 | 27 |
|------------------------------------------------------|-----|
| Subject Disposition: Informed Consent and Enrollment | |
| All Subjects | |
| Listing 16.2.1.2 | 28 |
| Inclusion/Exclusion Criteria Not Met | |
| All Subjects | |
| Listing 16.2.1.3 | 29 |
| Subject Disposition: End of Study | |
| All Dosed Subjects | |
| Listing 16.2.1.4 | 30 |
| Follow-Up Telephone Visit | |
| All Dosed Subjects | |
| Listing 16.2.2.1 | 31 |
| Protocol Deviations | |
| All Subjects | |
| Listing 16.2.4.1 | |
| Demographics | |
| All Subjects | |
| Listing 16.2.4.2 | |
| Cushing's Syndrome Medical History | |
| All Subjects | |
| Listing 16.2.4.3 | |
| Tobacco Use | |
| All Subjects | |
| Listing 16.2.4.4 | |
| General Medical History | |
| All Subjects | |
| Listing 16.2.4.5 | 36 |
| Pituitary Radiotherapy | |
| All Subjects | |
| Listing 16.2.4.6 | |
| Prior and Concomitant Medications | |
| All Subjects | |
| Listing 16.2.4.7 | 38 |
| Concomitant Procedures | |
| All Subjects | 26 |
| Listing 16.2.5.1 | 39 |
| Study Drug Administration | |
| All Dosed Subjects | 4.6 |
| Listing 16.2.5.2 | 40 |
| Study Drug Accountability | |
| All Dosed Subjects | А 1 |
| Listing 16.2.5.3 | 41 |
| Study Drug Exposure and Compliance | |
| All Dosed Subjects | |

| Listing 16.2.6.1 | 42 |
|----------------------------------------------------------|----|
| 24 Hour Urine Laboratory Results | |
| All Subjects | |
| Listing 16.2.6.2 | 43 |
| ARUP Laboratories: Plasma and Serum Samples | |
| All Subjects | |
| Listing 16.2.6.3 | 44 |
| ARUP Laboratories: Urine Samples | |
| All Subjects | |
| Listing 16.2.6.4 | 45 |
| Salivary Cortisol | |
| All Subjects | |
| Listing 16.2.6.5 | 46 |
| Hormones | |
| All Subjects | |
| Listing 16.2.6.6 | 47 |
| Pharmacokinetic Samples | |
| All Dosed Subjects | |
| Listing 16.2.7.1 | 48 |
| Adverse Events | |
| All Subjects | |
| Listing 16.2.8.1 | 49 |
| Safety Laboratory Values: Chemistry | |
| All Subjects | |
| Listing 16.2.8.2 | 50 |
| Safety Laboratory Values: Hematology | |
| Screened Subjects | |
| Listing 16.2.8.3 | 50 |
| Safety Laboratory Values: Lipids | |
| Screened Subjects | |
| Listing 16.2.8.4 | 50 |
| Safety Laboratory Values: Coagulation | |
| Screened Subjects | |
| Listing 16.2.8.5 | 50 |
| Safety Laboratory Values: Urinalysis | |
| Screened Subjects | |
| Listing 16.2.8.6 | 50 |
| Safety Laboratory Values: Serology and Urine Drug Screen | |
| Screened Subjects | |
| Listing 16.2.8.7 | 51 |
| Serum and Urine Pregnancy Test | |
| All Subjects | |
| Listing 16.2.9.1 | 52 |
| Vital Signs | |
| All Subjects | |
| Listing 16.2.9.2 | 53 |

| 12-L | Lead Electrocardiogram | |
|---------|------------------------|----|
| All S | Subjects | |
| Listing | g 16.2.9.3 | 54 |
| | sical Examination | |
| All S | Subjects | |

## Listing 16.2.1.1 Subject Disposition: Informed Consent and Enrollment All Subjects

| Subject | Date of<br>Informed<br>Consent | Did Subject Enroll<br>In the Open-Label<br>Dose Escalation Period? | Date<br>Enrolled | Date of<br>Screen Failure | Reason for Screen Failure | Did Subject Continue to the<br>Double-Blind Randomized<br>Withdrawal Period or the<br>Additional Open-Label Dosing? |
|---|---|---|---|---|---|---|
| ###-### | DDMMMYYYY | YES | DDMMMYYYY | | | NO |
| ###-## | DDMMMYYYY | NO | | DDMMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| ###-### | DDMMMYYYY | YES | DDMMMYYYY | | | NO |
| ###-### | DDMMMYYYY | YES | DDMMMYYYY | | | NO |
| ###-## | DDMMMYYYY | YES | DDMMMYYYY | | | NO |
| ###-## | DDMMMYYYY | NO | | DDMMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |

<sup>&</sup>lt;< <u>Programming Note</u>: Refer to records where DS.DSDECOD = "INFORMED CONSENT OBTAINED", DS.DSSCAT = "ENROLLMENT", DS.DSSCAT = "SCREEN FAILURE", and DS.DSCAT = "PROTOCOL MILESTONE". >>

## Listing 16.2.1.2 Inclusion/Exclusion Criteria Not Met All Subjects

| Subject | Category | Criterion | Description |
|---|---|---|---|
| ###-### (SF) | xxxxxxxx | ## | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | xxxxxxxx | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-## | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### (SF) | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### (SF) | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### (SF) | XXXXXXXX | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-### (SF) | xxxxxxxx | ## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

SF = Screen failure subject

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Only use the last 2 digits of IE.IETESTCD for the criterion number. >>

# Listing 16.2.1.3 Subject Disposition: End of Study All Dosed Subjects

| Subject | Date of<br>First Dose | Date (Day) of<br>Last Dose | Completed<br>Study? | Date (Day) of<br>Completion/<br>Early Termination | Primary Reason for Early Termination |
|---|---|---|---|---|---|
| ###-##<br>###-##<br>###-##<br>###-## | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY (##) DDMMMYYYYY (##) DDMMMYYYYY (##) | XXX<br>XXX<br>XXX | DDMMMYYYY (##) DDMMMYYYYY (##) DDMMMYYYYY (##) DDMMMYYYYY (##) | ************************************** |

Day = Date - first dose date +1.

#### Listing 16.2.1.4 Follow-Up Telephone Visit All Dosed Subjects

| Subject | Was the Subject<br>Reached for<br>Follow-Up? | Date (Day)<br>of Contact | Any Adverse Events<br>Since Last<br>Study Visit? | Started or Stopped<br>Any Medications Since<br>Last Study Visit? |
|---|---|---|---|---|
| ###-### | XXX | DDMMMYYYY (##) | XXX | XXX |
| ###-### | XXX | DDMMMYYYY (##) | XXX | XXX |
| ###-## | XXX | DDMMMYYYY (##) | XXX | XXX |
| ###-### | XXX | DDMMMYYYY (##) | XXX | XXX |

Day = Date - first dose date +1.

Listing 16.2.2.1 Protocol Deviations All Subjects

| Subject | Date of<br>Verification | Date of<br>Occurrence | Pre-<br>Approved? | Category | Description | CSR<br>Reportable? | Action Type | Confirmed? |
|---|---|---|---|---|---|---|---|---|
| ###-## | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | xxxxxxxxxxxxxxx | XXX | xxxxxxxxxxxxxxxxxx | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXXX | xxxxxxxxxxxxxxxx | XXX | xxxxxxxxxxxxxxxxxx | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| ###-### (SF) | DDMMMYYYY | DDMMMYYYY | XXX | xxxxxxxxxx | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| , , | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | xxxxxxxxxxxxxxxxxx | XXX |
| ###-### | DDMMMYYYY | DDMMMYYYY | XXX | xxxxxxxxxx | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| ###-### | DDMMMYYYY | DDMMMYYYY | XXX | xxxxxxxxxx | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |
| | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXXXX | XXXXXXXXXXXXXXXX | XXX | XXXXXXXXXXXXXXXXXXXXXX | XXX |

SF = Screen failure subject. CSR = Clinical Study Report.

Listing 16.2.4.1 Demographics All Subjects

| Subject | Protocol<br>Version | Date of<br>Birth | Age<br>(Years) | Sex | Ethnicity | Race | Race, Specify |
|---|---|---|---|---|---|---|---|
| ###-## (SF) | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| ###-## | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## (SF) | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## (SF) | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## (SF) | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | XXXXXXXXX | DDMMMYYYY | ## | XXXX | XXXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXX |

SF = Screen failure subject

# Listing 16.2.4.2 Cushing's Syndrome Medical History All Subjects

| Subject | Diagnosis<br>Date | Etiology | How was the etiology confirmed? | History of Prior<br>Pituitary Surgery? | Previous Pituitary<br>Radiotherapy? |
|---|---|---|---|---|---|
| ###-### (SF) | DDMMMYYYY | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX | XXX |
| ###-## | DDMMMYYYY | XXXXXXXX | *************************************** | XXX | xxx |
| ###-### (SF) | DDMMMYYYY | XXXXXXXX | ************ | XXX | xxx |
| ###-### | DDMMMYYYY | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | xxx |
| ###-## | DDMMMYYYY | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | XXX |

SF = Screen failure subject

#### Listing 16.2.4.3 Tobacco Use All Subjects

| Subject | Cigarette Use | Frequency | Other Tobacco Product use |
|--------------|-----------------|----------------|---------------------------|
| ###-### (SF) | NEVER SMOKED | | NEVER USED |
| ###-## | FORMERLY SMOKED | xxxxxxxxxxxx | NEVER USED |
| ###-## | XXXXXXXXXXXXX | xxxxxxxxxxxx | xxxxxxxxx |
| ###-## | xxxxxxxxxxxx | XXXXXXXXXXXXXX | XXXXXXXXX |

SF = Screen failure subject

Program Name: XXXXXXXX.sas

Run Date: DDMMMYYYY HH:MM

Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: If other data is reported, e.g. number of cigarettes, other tobacco product information, or start/stop dates, then add columns for the additional data. >>

#### Listing 16.2.4.4 General Medical History All Subjects

| Subject | System Organ Class/<br>Preferred Term/<br>Event/Diagnosis | Start Date | Stop Date |
|---|---|---|---|
| ###-### (SF) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | ONGOING |
| ###-### | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |

SF = Screen failure subject. Medical history is coded using MedDRA dictionary version 18.0.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Only include records where MHPRESP=null. Sort by USUBJID, MHSTDTC, MHENDTC, MHTERM. >>

# Listing 16.2.4.5 Pituitary Radiotherapy All Subjects

| Subject | Date of First Dose | Date of Last Dose | Comments |
|---|---|---|---|
| ###-## | DDMMMYYYY | DDMMMYYYY | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| Program Name: XXXXXXXX.sas | | Run Date: DDMMMYYYY HE | 1:MM Clinical database last extracted: DDMMYYYY HH:MM |
## Listing 16.2.4.6 Prior and Concomitant Medications All Subjects

| Subject | Medication Name/<br>Preferred Term/<br>Chemical Substance | Start Date/<br>End Date | Indication | Dose | Units | Frequency | Route |
|---|---|---|---|---|---|---|---|
| ###-### | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>DDMMMYYYY | xxxxxxxxxxxxx | xxxxxx | XXXXX | OTHER: XXXXXXX | xxxxxxxxxx |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>ONGOING | xxxxxxxxxxxxxx | XXXXXXX | OTHER:<br>XXXXXXXXX | XXXXXXXXX | xxxxxxxxx |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>ONGOING | xxxxxxxxxxxxxx | XXXXXXX | XXXXX | XXXXXXXXX | OTHER: XXXXXXXXX |
| ###-## | xxxxxxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxx | DDMMMYYYY/<br>DDMMMYYYY | xxxxxxxxxxxxxxx | XXXXXXX | XXXXX | XXXXXXXXX | xxxxxxxxxx |
| ###-### | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXXXXXXXXXXXXX | XXXXXXX | XXXXX | XXXXXXXXX | xxxxxxxxxx |

Medications are coded with the WHO Drug March 2016E B2 dictionary version.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Sort by USUBJID, CMSTDTC, CMENDTC, CMTRT. >>

Program Name: XXXXXXXX.sas

#### Listing 16.2.4.7 Concomitant Procedures All Subjects

| Subject | Procedure | Indication | Start Date | Stop Date |
|---|---|---|---|---|
| ###-## | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | xxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxx | DDMMMYYYY | ONGOING |
| ###-## | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxx | DDMMMYYYY | DDMMMYYYY |
| ###-## | xxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxx | DDMMMYYYY | DDMMMYYYY |
| ###-### | xxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |

Run Date: DDMMMYYYY HH:MM

Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Sort by USUBJID, PRSTDTC, PRENDTC, PRTRT. >>

#### Listing 16.2.5.1 Study Drug Administration All Dosed Subjects

| Subject | Visit | Treatment Name | Date/Time of<br>Administration | Did Subject Consume<br>Food Prior to<br>Administration? | Was the Planned Dose<br>Administered On Site? |
|---|---|---|---|---|---|
| ###-### | xxxxxxxxxxx | Nevanimibe 250 mg BID | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | Nevanimibe 500 mg BID | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | Nevanimibe 1000 mg BID | DDMMMYYYY/HH:MM | XXX | XXX |
| ###-## | XXXXXXXXXXX | xxxxxxxxxxxx | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| ###-## | XXXXXXXXXXX | xxxxxxxxxxxx | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| ###-### | XXXXXXXXXXX | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| | XXXXXXXXXXX | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXX | XXX |
| | | | , . | | |

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: Only include records where ECOCCUR = "Y". >>

#### Listing 16.2.5.2 Study Drug Accountability All Dosed Subjects

| | | Treatment | Disp | Dispense | | urn | |
|---|---|---|---|---|---|---|---|
| Subject | Bottle<br>Number | | Date | Number of<br>Tablets | Date | Number of<br>Tablets | 80-120%<br>Compliant? |
| ###-### | #####<br>#####<br>##### | Nevanimibe 250 mg BID<br>Nevanimibe 500 mg BID<br>Nevanimibe 1000 mg BID<br>Nevanimibe 1000 mg BID | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | # #<br># #<br># #<br># # | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | # #<br># #<br># # | XXX<br>XXX<br>XXX<br>XXX |
| ###-### | #####<br>#####<br>##### | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | ##<br>##<br>## | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | # #<br># #<br># # | XXX<br>XXX<br>XXX |

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

 $<< \underline{Programming\ Note}:$  Sort by Subject, Dispense Date, Return Date. The compliance question is sourced from SUPPDA where QNAM = "COMP".>>

#### Listing 16.2.5.3 Study Drug Exposure and Compliance All Dosed Subjects

| | Nevanimibe 250 mg BID | | Nevanimibe 500 mg BID | | | Nevanimibe 1000 mg BID | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Number of<br>Tablets | Days of<br>Exposure | Compliance<br>(%) | Number of<br>Tablets | Days of<br>Exposure | Compliance | Number of<br>Tablets | Days of<br>Exposure | Compliance |
| ###-## | ## | ## | ###.# | ## | ## | ###.# | ## | ## | ###.# |
| ###-## | ## | ## | ###.# | ## | ## | ###.# | | | |
| ###-## | ## | ## | ###.# | ## | ## | ###.# | ## | ## | ###.# |
| ###-## | ## | ## | ###.# | ## | ## | ###.# | ## | ## | ###.# |

Number of tablets = number of tablets dispensed - number of tablets returned.

Days of exposure = last dose date of the specified dose level - first dose date of the specified dose level +1.

Compliance = 100\*number of tablets/(days of exposure\*2) for the 250 mg BID and 500 mg BID groups.

Compliance = 100\*number of tablets/(days of exposure\*4) for the 1000 mg BID group.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: For the last dose level (i.e. 500 mg for subject 103-001 and 1000 mg for others), exposure = TRTEDT – TR03SDT + 1. For other dose levels, assume that the "last dose date of the specified dose level" is the day before the first dose date of the next dose level. For example for 250 mg (except 103-001), exposure = TR02SDT – TR01SDT. >>

## Listing 16.2.6.1 24 Hour Urine Laboratory Results All Subjects

| Subject | Parameter (Unit) | Visit | Collection Start<br>Date/Time | Collection End<br>Date/Time | Result | Normal Range | Flag |
|---|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXX (XXXXX) | xxxxxxxxxx | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | xx - xx | |
| """ (02) | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | HIGH |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | 112 011 |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | LOW |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | xx - xx | |
| | , | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-## | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-## | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | xx - xx | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: Include all results where LBCAT = "24 HOUR URINE".

In all lab listings, report results in US conventional units (LBORRES variables). >>

## Listing 16.2.6.2 ARUP Laboratories: Plasma and Serum Samples All Subjects

| Subject | Parameter (Unit) | Visit | Date/Time of<br>Collection | Result | Normal Range | Flag |
|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | HIGH |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | LOW |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-## | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-### | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | . , | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Include all results where LBCAT = "ARUP LABORATORIES" and LBSPEC in ("PLASMA", "SERUM")>>

<< <u>Programming Note</u>: The following will have the same layout as listing 16.2.6.1. Include all results where LBCAT = "ARUP LABORATORIES" and LBSPEC = "URINE". >>

Listing 16.2.6.3
ARUP Laboratories: Urine Samples
All Subjects

Listing 16.2.6.4 Salivary Cortisol All Subjects

| Subject | Parameter (Unit) | Visit | Time Point | Date/Time of<br>Collection | Result | Normal Range | Flag |
|---|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | xx - xx | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | HIGH |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | LOW |
| | | XXXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | xxxxxxxxxxx | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-### | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | xxxxxxxxxxx | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| ###-### | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | , , | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |
| | | XXXXXXXXXXX | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<< <u>Programming Note</u>: Include all results where LBSPEC = "SALIVA" (includes LBCAT = "HORMONES" and "ARUP LABORATORIES"). >>

<< <u>Programming Note</u>: I am waiting to see how the salivary cortisol collection CRFs are mapped to see how best to list the data  $(SC1 = questions \ about \ shift \ work, \ travel, \ altered \ wake/sleep \ and \ LB\_SC1 = smoking \ question) >>$ 

<< <u>Programming Note</u>: The following will have the same layout as listing 16.2.6.2. Include all results where LBCAT in("HORMONES", "QUEST DIAGNOSTICS") and LBSPEC NE "SALIVA". >>

Listing 16.2.6.5 Hormones All Subjects Program Name: XXXXXXXX.sas

Clinical database last extracted: DDMMYYYY HH:MM

## Listing 16.2.6.6 Pharmacokinetic Samples All Dosed Subjects

| Subject<br>Visit | Last Dose Prior<br>to PK Sampling<br>Date/Time | Sampling<br>Time Point | Date/Time | Nevanimibe (< <unit>&gt;)</unit> | If Not Collected,<br>Specify Reason |
|---|---|---|---|---|---|
| # # # <b>-</b> # # # | | | | | |
| XXXXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| XXXXXXXXXXXXXX | | | NOT DONE | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| | | XXXXXXXXXX | DDMMMYYYY/HH:MM | ###### | |
| XXXXXXXXXXXXXX | | | NOT DONE | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

<< <u>Programming Note</u>: Include footnotes for the lower limits of quantitation if provided. Include columns for each metabolite provided, delete if not needed. >>

Run Date: DDMMMYYYY HH:MM

#### Listing 16.2.7.1 Adverse Events All Subjects

| Subject | | Adverse Event/<br>Preferred Term/<br>System Organ Class | Start Date/Day<br>End Date/Day | Duration<br>(Days) | Severity/<br>Relationship<br>to Study Drug | Action Taken<br>with Study Drug | Outcome/<br>Other Action Taken |
|---|---|---|---|---|---|---|---|
| ###-### | YES/<br>250 mg/<br>NO | XXXXXXXXXXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXX | DDMMMYYYY/##<br>DDMMMYYYY/## | ## | XXXXXX/<br>XXXXXXXXXXXX | DOSE NOT CHANGED | xxxxxxx/<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | YES/<br>1000 mg/<br>XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/##<br>DDMMMYYYY/## | ## | XXXXXX/<br>XXXXXXXXXXXX | DRUG INTERRUPTED Last Dose: DDMMMYYYY Restart: DDMMMYYYY | XXXXXXX/<br>XXXXXXXXXXXXXX |
| ###-### | NO/<br>Pre-dose/<br>XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/##<br>DDMMMYYYY/## | ## | XXXXXX/<br>XXXXXXXXXXXX | xxxxxxxxxxx | xxxxxxx/<br>xxxxxxxxxxxxxxxx |
| ###-### | YES/<br>500 mg/<br>XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/##<br>DDMMMYYYY/## | ## | XXXXXX/<br>XXXXXXXXXXX | xxxxxxxxxxx | xxxxxxx/<br>xxxxxxxxxxxxxxx |

TEAEs are defined as any AE beginning on or after the first dose date of study drug. Onset dose is the subject's Nevanimibe dose level on the reported start date of the event. For AEs starting prior to first dose of study drug, day = start date/end date - first dose of study drug. Otherwise, day = start date/end date - first dose date OF THE ONSET DOSE LEVEL +1. Duration = end date - start date + 1.

AEs are coded using MedDRA dictionary version 18.0.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Refer to EC.ECCAT="EXCEPTION DOSE" for the date of last dose prior to interruption and the date of restart. If any additional free text is mapped to SUPPAE (e.g. outcome sequelae or specify other action taken), then list it with the text of the parent field. >>

Millendo Therapeutics US, Inc. Protocol ATR-101-301

Page 1 of #

## Listing 16.2.8.1 Safety Laboratory Values: Chemistry All Subjects

| Subject | Parameter (Unit) | Visit | Date/Time of<br>Collection | Result | Normal Range | Flag [1] |
|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXX (XXXXX) | xxxxxxxxxxx | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| (, | (, | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | XXXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| ###-## | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| ###-## | XXXXXXXXXX (XXXXX) | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |
| | | XXXXXXXXXXX | DDMMMYYYY/HH:MM | XXXXX | XX - XX | XX |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

<sup>[1]</sup> Laboratory Flag: RH=Reference High, RL=Reference Low, NH=Notable High, NL=Notable Low, CH=Critical High, CL=Critical Low

<sup>&</sup>lt;< <u>Programming Note</u>: Including all non-missing LBORRES where LBCAT = "CHEMISTRY". Exclude LBTESTCD = "HCG" since that is a pregnancy test which is included in another listing. >>

#### <u>Programming Note</u>: The following listings will have the same layout as Listing 16.2.8.1.

Listing 16.2.8.2
Safety Laboratory Values: Hematology
Screened Subjects

Listing 16.2.8.3
Safety Laboratory Values: Lipids
Screened Subjects

Listing 16.2.8.4
Safety Laboratory Values: Coagulation
Screened Subjects

Listing 16.2.8.5
Safety Laboratory Values: Urinalysis
Screened Subjects

Listing 16.2.8.6
Safety Laboratory Values: Serology and Urine Drug Screen
Screened Subjects

## Listing 16.2.8.7 Serum and Urine Pregnancy Test All Subjects

| Subject | Visit | Date of Last<br>Menstrual Period | Collection<br>Date/Time | Urine Test<br>Result | Serum Test<br>Result | Reason Not Done |
|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXXXXX<br>XXXXXXXXXXXXX<br>XXXXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY/HH:MM DDMMMYYYY/HH:MM DDMMMYYYY/HH:MM DDMMMYYYY/HH:MM | XXXXXXX<br>XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXX | ************************************** |
| ###-### | XXXXXXXXXXXX<br>XXXXXXXXXXXXX<br>XXXXXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY/HH:MM DDMMMYYYY/HH:MM DDMMMYYYY/HH:MM DDMMYYYYY/HH:MM DDMMYYYYY/HH:MM | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | ************************************** | ************************************** |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

<< <u>Programming Note</u>: Include all records where LB.LBTESTCD = "HCG" and LBNAM = null. >>

Listing 16.2.9.1 Vital Signs All Subjects

| Subject | Visit | Date<br>Performed | SBP<br>(mmHg) | DBP<br>(mmHg) | HR<br>(bpm) | Temperature<br>(Units) | RR<br>(bpm) | Weight<br>(Units) | Height<br>(Units) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°C) | ### | ###.# (lb) | ###.# (in) | ##.# |
| ###-### | xxxxxxxxxxx | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°C) | ### | ###.# (lb) | ###.# (in) | ##.# |
| ###-## | xxxxxxxxxxx | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°F) | ### | ###.# (kg) | ###.# (cm) | ##.# |
| | XXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### (°C) | ### | ###.# (lb) | ###.# (in) | ##.# |

SF = Screen failure subject.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYY HH:MM

SBP = systolic blood pressure. DBP = diastolic blood pressure. HR = heart rate (bpm = beats per minute).

RR = respiratory rate (bpm = breaths per minute). BMI = Body Mass Index.

#### Listing 16.2.9.2 12-Lead Electrocardiogram All Subjects

| Subject<br>Visit | Date<br>Performed | Heart Rate (beats/min) | <br>PR | · Inte<br>QRS | erval<br>QT | (msec)<br>QTcF | RR | Overall Interpretation | Describe Abnormality |
|---|---|---|---|---|---|---|---|---|---|
| ###-### (SF) | | | | | | | | | |
| XXXXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | NORMAL | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | ABNORMAL, NCS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | ABNORMAL, CS | XXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | XXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | | | | | | | | | |
| XXXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | XXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | XXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | XXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXXXXXXXX | DDMMMYYYY | ### | ### | ### | ### | ### | ### | XXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

SF = Screen failure subject. NCS = not clinically significant. CS = clinically significant.

Program Name: XXXXXXXX.sas Run Date: DDMMYYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM

# Listing 16.2.9.3 Physical Examination All Subjects

| Subject | Visit | Date of Exam | Result | Describe Findings |
|---|---|---|---|---|
| ###-### (SF) | XXXXXXXXXXXXXX | DDMMMYYYY | NORMAL | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | ABNORMAL NCS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | NO CHANGE FROM PREVIOUS EXAM | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | ABNORMAL CS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ###-## | XXXXXXXXXXXXXX | DDMMMYYYY | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXX | DDMMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

 ${\tt SF} = {\tt Screen}$  failure subject.  ${\tt CS} = {\tt Clinically}$  significant.  ${\tt NCS} = {\tt Not}$  clinically significant.

Program Name: XXXXXXXX.sas Run Date: DDMMMYYYY HH:MM Clinical database last extracted: DDMMYYYYY HH:MM